CLINICAL TRIAL: NCT01349712
Title: Correlation of Feasibility Batches Using Warfarinised Blood
Brief Title: Study to Test the Accuracy of a Prototype Handheld PT/INR Device
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Universal Biosensors Pty Ltd (Industry)
Responsible Party: Richard Ward, Assistant Professor, College of Pharmacy Harding University
Other Study IDs: MOB 0158
Record Dates: First submitted 2011-04-29; First posted 2011-05-09 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2011-05

CONDITIONS: Blood Coagulation Disorders
MeSH Terms: conditions — Blood Coagulation Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Coumadin (warfarin): Subjects are required to be currently receiving coumadin (warfarin) treatment.

SUMMARY:
The purpose of this study is to measure prothrombin time (PT) on an experimental device and a commercially available device on persons receiving coumadin (warfarin)treatment.

DETAILED DESCRIPTION:
This study will require participants to have up to 2 finger-punctures taken and sample tested on a strip and meter system for both the experimental and commercially available devices.

ELIGIBILITY:
Inclusion Criteria:

* Currently taking coumadin (warfarin)
* Aged 18 years or older
* Able and willing to provide informed consent
* Can understand (read and write) English

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects currently receving coumadin(warfarin) treatment
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
PT/INR values from the experimental device will be statistically correlated to results obtained from a commercially available device | Fives days to collect data and up to two weeks to generate correlation graph
  To determine the correlation of PT/INR values between an experimental and commercial device.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Ward, Pharm D, Principal Investigator — Harding University
Locations (1):
- White River Diagnostic Clinic, Batesville, Arkansas, United States